CLINICAL TRIAL: NCT04125212
Title: Effects of Air Pollution on Cardio-metabolic Outcomes Among Heathy Adults
Brief Title: Air Pollution and Cardio-metabolic Health
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University (Other)
Responsible Party: Principal Investigator, WeiHuang, Principal Investigator, Peking University
Other Study IDs: WeiHuang
Record Dates: First submitted 2019-10-11; First posted 2019-10-14 (Actual); Last update posted 2021-09-16 (Actual); Status verified 2021-09

CONDITIONS: Cardiovascular Outcomes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Collection of blood and urine samples
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
To investigate the effects of air pollution on surrogate cardio-metabolic outcomes in young healthy adults.

DETAILED DESCRIPTION:
To investigate the effects of air pollution on surrogate cardio-metabolic outcomes in a panel study involving young healthy adults living in Beijing, China with extreme high ambient air pollution levels.

ELIGIBILITY:
Inclusion Criteria:

1. Living in Peking University Health Science Center neighborhood.
2. Non smoker and no diseases.

Exclusion Criteria:

1. Advanced microvascular complications and active cardiovascular disease.
2. Pregnancy or intent to get pregnant during the study period.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: non-smoker young healthy adults
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2019-09-21 (Actual); Primary Completion 2020-01-16 (Actual); Study Completion 2022-06-01 (Estimated)

PRIMARY OUTCOMES:
Blood pressure | Four months
  Systolic blood pressure and diastolic blood pressure

SECONDARY OUTCOMES:
Systemic inflammatory | Four months
  Systemic inflammation biomarkers, such as C-reactive protein etc.

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University ,School of Public Health, Beijing, Beijing Municipality, China